CLINICAL TRIAL: NCT00818584
Title: A Phase 1 Open-Label Study of the Safety and Pharmacokinetics of Repeated-Dose Micafungin in Neonates
Brief Title: An Open-Label Study of the Safety and Pharmacokinetics of Repeated-Dose Micafungin in Neonates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 9463-CL-2104; NCT00906230 (obsolete NCT alias)
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Candida
Keywords: Micafungin; Candida; Neonates; Mycamine; FK463
MeSH Terms: conditions — Torulopsis | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. micafungin lower dose (Experimental)
  Interventions: Drug: Micafungin
- 2. micafungin higher dose (Experimental)
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — IV Administration
  Other Names: Mycamine; FK463

SUMMARY:
This study will evaluate pharmacokinetics and safety of intravenous micafungin in neonates with suspected candida infection

DETAILED DESCRIPTION:
Subjects will be stratified by weight to receive one of two doses of study drug

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and HIPAA authorization of the infant's parent or legally authorized representative must be obtained prior to study entry
* Infant has sufficient venous access to permit study drug dosing
* Infant is suspected to have a systemic Candida infection and appropriate cultures (blood with or without urine/CSF) are obtained at the time of study entry

Exclusion Criteria:

* Infant has a history of anaphylaxis, hypersensitivity, or any serious reaction to the echinocandin class of antifungals
* Infant has received an echinocandin within one month prior to study entry
* Infant has a concomitant medical condition which, in the opinion of the investigator and/or medical advisor, may create an unacceptable additional risk
* Infant has a life expectancy of less than 96 hours

Ages: 48 Hours to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Assessment of micafungin plasma pharmacokinetic parameters | Day 4

SECONDARY OUTCOMES:
Monitor adverse events | 11 or 12 Days

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (7):
- United States (7):
  - Birmingham, Alabama
  - Orange, California
  - Louisville, Kentucky
  - Kansas City, Missouri
  - Durham, North Carolina
  - Dallas, Texas
  - Charlottesville, Virginia

REFERENCES:
- [Background] Benjamin DK Jr, Smith PB, Arrieta A, Castro L, Sanchez PJ, Kaufman D, Arnold LJ, Kovanda LL, Sawamoto T, Buell DN, Hope WW, Walsh TJ. Safety and pharmacokinetics of repeat-dose micafungin in young infants. Clin Pharmacol Ther. 2010 Jan;87(1):93-9. doi: 10.1038/clpt.2009.200. Epub 2009 Nov 4. PMID 19890251